CLINICAL TRIAL: NCT04604223
Title: Effect of Pioglitazone on Inflammatory Response and Clinical Outcome in T2DM Patients With COVID-19
Brief Title: Effect of Pioglitazone on T2DM Patients With COVID-19
Acronym: PIOQ8
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dasman Diabetes Institute (Other)
Collaborators: Ministry of Health, Kuwait (Other Government); Texas Diabetes Institute (Other); Kuwait University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RA HM-2020- 011
Record Dates: First submitted 2020-10-26; First posted 2020-10-27 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2020-10

CONDITIONS: Covid19; Type 2 Diabetes
MeSH Terms: conditions — COVID-19; Diabetes Mellitus, Type 2 | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pioglitazone (Experimental): Pioglitazone will be started at 45 mg/day dose for 10 days, after 10 days, the dose will be reduced to 30 mg/day to minimize possible adverse events. The treatment will be continued for 4 weeks (28 days) total.
  Interventions: Drug: Pioglitazone 45 mg
- Placebo (Placebo Comparator): Placebo tablets at 45 mg/day will be given for 10 days, after 10 days, the tablets will be reduced to 30 mg/day. The treatment will be continued for 4 weeks (28 days) total.
  Interventions: Drug: Pioglitazone 45 mg

INTERVENTIONS:
Drug: Pioglitazone 45 mg — Pioglitazone will be started at 45 mg/day dose for 10 days, after 10 days, the dose will be reduced to 30 mg/day to minimize possible adverse events. The treatment will be continued for 4 weeks (28 days) total

SUMMARY:
Approximately 10-15% of patients infected with COVID-19 develop severe illness characterized by respiratory distress, increased risk of clotting disease, myocardial damage, stroke and mortality. Subjects with Type 2 diabetes (T2DM) are at increased risk for severe COVID-19 disease. Exuberant inflammatory and immune responses were suggested as the etiology responsible for the development of severe COVID-19 disease. The increased chronic inflammatory state characteristic of T2DM could contribute to the increased risk of severe COVID-19 disease in T2DM patients. Therefore, its possible that anti-inflammatory therapy will reduce the risk of severe COVID-19 disease. Consistent with this assumption, a recent study has reported that steroid therapy improves the outcome in patients with severe COVID-19 disease.

The medication pioglitazone is a strong insulin sensitizer that reduces plasma glucose concentrations in T2DM patients. In addition to improving insulin sensitivity, several studies have demonstrated that pioglitazone reduces chronic inflammation in T2DM patients, which is manifested in a decrease in TNF-alpha, interleukin, hs CRP, leptin and other inflammatory markers in T2DM treated with pioglitazone. Further, pioglitazone enhances the plasma level of anti-inflammatory agents. For example, the plasma level of 15-epi-lipoxin A, a lipid mediator with strong anti-inflammatory and inflammation-resolving effects that has been reported to neutralize RNA coated viruses, is significantly elevated by pioglitazone treatment in T2DM patients. Therefore, we hypothesize that administering pioglitazone to T2DM patients who have moderate-to-severe COVID-19 will improve the clinical outcome of their COVID-19 disease.

DETAILED DESCRIPTION:
The study design is prospective, double blind, placebo-controlled trial aims to examine the effect of pioglitazone on inflammatory markers and clinical outcome in T2DM patients infected with COVID-19. 1506 T2DM patients with proven COVID-19 infection (positive swab) and at least one COVID-19 symptom will be randomized to receive in a double blind fashion pioglitazone or placebo for 28 days. Inflammatory response and a composite of clinical outcome will be measured at 3, 7, 14, 21 and 28 days (or time of discharge) after initiating therapy.

Study Design

1. Upon admission, subjects will be evaluated for inclusion and exclusion criteria. Eligible subjects will be consented.
2. After consenting, medical history and vital signs will be done including ECG and chest X-ray.
3. Blood for the following parameters (Panel 1, which are routinely measured for the management of COVID-19 patients) will be sent for measurement in the clinical lab: CBC, Full chemistry panel including LFT and RFT, lipid profile, blood gases, HbA1c, hsCRP, Troponin I, coagulation screen, D-Dimers, and Ferritin.

Study Intervention:

After completing baseline studies, subjects will be randomized in a double-blind fashion to receive: (1) pioglitazone, or (2) placebo. The study intervention will be introduced every morning at the same time for 4 weeks.

Because previous studies from Kuwait demonstrated that the mean hospitalization period for COVID-19 patients in Al-Jaber hospitals is 24 days.

Patient will be randomized based upon the following parameters: age, gender, BMI, baseline medications, background health conditions, diabetes duration, and respiratory rate. Each parameter will be monitored amongst both groups and the distribution of patients according to each parameter will be evenly distributed amongst the two treatment groups.

Pioglitazone will be started at 45 mg/day dose for 10 days, after 10 days, the dose will be reduced to 30 mg/day to minimize possible adverse events. The treatment will be continued for 4 weeks (28 days) total.

If during hospitalization, patient condition requires admission to ICU, respiratory support, or develops an increase in plasma troponin I levels (incidence of primary outcomes), pioglitazone/placebo therapy will be continued for the entire 4 weeks. Patient outcome will be evaluated weekly until end of week 4.

If patient condition is improved and patients is eligible for discharge (become asymptomatic plus O2 saturation >94% on room air) and he is discharged home prior to 4 weeks, blood tests will be drawn on discharge day, and patient will continue therapy at home to complete 4 week treatment period. At 28 days, a phone visit will be made to check on patient outcome. If discharged patients is readmitted due to deterioration in his clinical condition, the 28 day count will be considered since randomization.

Concomitant COVID-19 Therapy

1. Patients will receive standard of care for COVID-19 disease according to local guidelines. Other anti-inflammatory therapy or antiviral therapy for COVID-19 used in the medical center will be introduced to all patients unless prohibited by exclusion criteria. Reason for administration, administration dose, start date and duration of all medications introduced during hospitalization for COVID-19 therapy will be recorded.
2. Therapy for other background patient condition, e.g. blood pressure, cholesterol, etc. will be continued as per local guidelines.
3. If patient clinical condition through hospitalization precludes the use of pioglitazone (primarily due to fluid retention), the study intervention will be discontinued and distally acting diuretics (Aldactone 25 mg/day) will be started to reverse fluid retention.
4. If patient is transferred to other medical facility due to space issues (eg. transfer to field hospital), the patient will continue to be enrolled in the study, will receive study intervention and followed according to protocol in the other medical facility until discharge from the other medical facility.

Study End The study will end at end of week 4. Patients will be evaluated at end of week 4, and end of study data collection will be done, after which study intervention will be discontinued.

Measurement of compliance:

Study intervention will be administered in hospitalized patients or patients at other medical facilities under the supervision of medical team. If patients are discharged, they will continue therapy at home to complete the 4-week treatment period. Discharged patients will return to end of study visit at week 4, pill count will be performed at study end visit to evaluate patient compliance.

Glucose Control:

After completing the medical history, physical examination, and blood draws, if the patient receives SGLT2 inhibitor or metformin as antihyperglycemic therapy, they will be discontinued to reduce the risk of ketoacidosis and lactic acidosis, respectively. Sulfonylurea also will be discontinued to reduce the risk of hypoglycemia.

Patients who are not taking insulin for their antihyperglycemic therapy will be started on insulin. (see instructions below Table 1). Subjects receiving insulin therapy, if they receive basal/bolus insulin, the insulin dose will be adjusted to achieve the glucose treatment goals (140-180 mg/dl, 7.8-10 mM). subjects receiving premixed insulin will be switched to basal/bolus insulin as described below.

Daily blood glucose values will be measured every morning and according to local glucose monitoring policy according to patient needs.

Table 1: Instructions for starting insulin therapy

1. Discontinue oral antidiabetic drugs (sulfonylureas, repaglinide, nateglinide, metformin, SGLT2 inhibitors) on admission. Patients receiving DPP-4 inhibitors or GLP-1 RA will be allowed to continue these agents according to the treating physician discretion.
2. Starting insulin total daily dose (TDD): 0.5 units per kg of body weight. If patient is ≥ 70 years of age and/or with a serum creatinine ≥ 176 umol/l, reduce insulin TDD to 0.3 units per kg of body weight
3. Give half of total daily dose as insulin glargine and half as preprandial insulin
4. Administer insulin glargine once daily, at the same time of the day every day
5. Administer preprandial insulin in three equally divided doses before each meal.
6. If patient is unable to eat, hold the preprandial insulin
7. If patient receives GLP-1 RA as part of his diabetes management and you decide to continue GLP-1 RA therapy, hold the preprandial insulin
8. Adjust the glargine dose and preprandial insulin based upon the daily measured blood glucose levels to achieve a plasma glucose concentration 140-180 mg/dl (7.8-10 mM).
9. If patient's clinical condition requires admission to ICU, continues intravenous insulin infusion according to the protocol routinely used in the ICU is advised.

Other chronic diseases, including blood pressure, heart disease, lung disease, and all other medical conditions will be treated according to local guidelines or local treatment protocols for COVID-19 patients.

In hospital Follow-up:

Consistent with in patient care, daily medical history and physical examination will be done. The following parameters will be daily measured:

1. Mental status
2. Fever
3. Respiratory rate and use of auxiliary muscles
4. Oxygen saturation at room air or volume of oxygen flow rate needed to maintain oxygen saturation >95% (in patients without mechanical ventilation)
5. Heart rate and rhythm
6. Blood pressure Blood glucose levels will be measured according to hospital policy and insulin dose is adjusted to maintain blood glucose levels at the treatment range (140-180 mg/dl, 7.8-10 mM).

A complete follow-up visit with blood tests will be done at day 3,7, 14, 21, and 28.

All baseline Blood samples (Panel 1 and Panel 2) will be repeated at each follow-up visit. If patient clinical conditions are improved and the caring physician decided to discharge the patient home before the end of the week, all repeat blood samples will be done prior to discharge even if previous blood sample was less than one week. If patient will be transferred to a different medical facility or hospital to continue medical care, blood sample collection will be continued until patient is no longer part of the research protocol.

Criteria for discontinuation of study intervention:

The study intervention will be discontinued if:

1. Allergy to the study drug develops
2. Development of pulmonary congestion (based upon chest X-ray) requiring diuretic therapy
3. Peripheral edema requiring diuretic therapy
4. Withdraw consent

ELIGIBILITY:
Inclusion Criteria:

1. T2DM according to the ADA criteria. Patients with long standing diabetes as well as patients with new onset diabetes will be recruited. Patients receiving glucocorticoids for treatment of COVID-19 and manifest plasma glucose levels consistent with diabetes diagnosis also will be included
2. Patients can be drug naïve, receiving oral antihyperglycemic therapy (except pioglitazone), GLP-1 RA or insulin therapy will be allowed to participate in the study
3. COVID-19 infection confirmed with PCR test
4. Age 21-85 years
5. Patients of both sexes will be included
6. In addition to diabetes and COVID-19 diagnoses, patients should manifest at least one of COVID-19 symptoms (Fever, Chills, Headache, Rhinorreah, Cough (dry or with sputum), Sore Throat, shortness of breath, Hemoptysis, Altered mentation, Fatigue/Malaise, Myalgia, Nausea/Vomiting, Diarrhea, Anosmia, Chest pain).
7. Patient receiving other anti-inflammatory therapy for their routine COVID-19 care (e.g. hydroxychloroquine), or antiviral therapy (e.g. remdesivire) will be included in the study and will be evenly randomized amongst the two treatment groups

Exclusion Criteria:

1. T1DM
2. Absence of confirmation of COVID-19 infection
3. Age <21 years
4. Presence of heart failure (LVEF<40%) or a history of hospitalization for heart failure
5. Use of diuretics (furosemide or aldactone) for heart disease usually for heart failure. Patients with hypertension receiving diuretic therapy (usually thiazide) will be included in the study
6. Patient on mechanical ventilation or patients whose clinical condition requires mechanical ventilation in the following 24 hours.
7. Patients not expected to survive > 48 hours
8. Patients receiving pioglitazone for the management of their diabetes
9. Patients participating in other research study will be excluded
10. Pregnant women will be excluded from the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1506 (Estimated)
Dates: Start 2021-01-18 (Actual); Primary Completion 2021-06-29 (Estimated); Study Completion 2021-06-29 (Estimated)

PRIMARY OUTCOMES:
HsCRP level | 4 weeks
  Difference from baseline to 4 weeks in inflammatory response between subjects receiving pioglitazone versus placebo measured as plasma hsCRP level.
Difference in the incidence at 4 weeks of a composite outcome comprised of: | 4 weeks
  1) requirement for mechanical ventilation (invasive [with tracheal tube] or non-invasive); 2) myocardial damage measured as plasma troponin I level > 3 times the upper normal limit; or 3) death.

SECONDARY OUTCOMES:
Number of days free of mechanical ventilation | 4 weeks
Number of days in the ICU | 4 weeks
Duration of hospitalization | 4 weeks
Change from baseline in qSOFA score | 4 Weeks
Change from baseline in SO2/FiO2 | 4 Weeks
Difference in respiratory rate | 4 weeks
  Difference in respiratory rate, measured as the area under the curve of respiratory rate over time from baseline to week 4
Incidence at 4 weeks of a composite of extrapulmonary disease comprised of : | 4 weeks
  (a) myocardial disease measured as troponin I above the normal limit at any time during hospitalization, (b) neurologic disease manifested as TIA, or symptoms of peripheral or central neurologic deficient at anytime during hospitalization, (c) renal failure measured as > 50% decrease in eGFR

CONTACTS AND LOCATIONS:
Overall Officials: Fahd Al-Mulla, PhD, Principal Investigator — Dasman Diabetes Institute; Thamer Alessa, MD, Principal Investigator — Dasman Diabetes Institute. Ministry of Health, Kuwait; Mohamed Abu-farha, Principal Investigator — Dasman Diabetes Institute; Muhammed Abdul-Ghani, MD/PhD, Principal Investigator — Texas Diabetes Institute
Locations (5):
- Kuwait (4):
  - Al-Amiri Hospital, Kuwait City, (Pick From List)
  - Jaber Al Ahmad Al Sabah Hospital, Kuwait City, (Pick From List)
  - Mishrif Field Hospital, Kuwait City, (Pick From List)
  - Mubarak Al-Kabeer Hospital, Kuwait City, (Pick From List)
- Hamad Medical Corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baagar K, Alessa T, Abu-Farha M, Abubaker J, Alhumaidi H, Franco Ceruto JA, Hamad MK, Omrani A, Abdelrahman S, Zaka-Ul Haq M, Safi AW, Alhariri B, Barman M, Abdelmajid A, Cancio HVD, Elmekaty E, Al-Khairi I, Cherian P, Jayyousi L, Ahmed M, Qaddoumi M, Hajji S, Esmaeel A, Al-Andaleeb A, Channanath A, Devarajan S, Ali H, Thanaraj TA, Al-Sabah S, Al-Mulla F, Abdul-Ghani M, Jayyousi A. Effect of pioglitazone on inflammatory response and clinical outcome in T2DM patients with COVID-19: a randomized multicenter double-blind clinical trial. Front Immunol. 2024 Sep 6;15:1369918. doi: 10.3389/fimmu.2024.1369918. eCollection 2024. PMID 39308871